CLINICAL TRIAL: NCT06467032
Title: Evaluation of the Effectiveness and Tolerance of Cicaplast Baume B5 on the Re-epithelialization Kinetic After Superficial CO2 Laser Resurfacing
Brief Title: Effectiveness and Tolerance of Cicaplast Baume B5 After Superficial CO2 Laser Resurfacing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LRP21007 Cicaplast
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Wound Heal
Keywords: re-epithelialization; superficial CO2 laser resurfacing; Cicaplast Baume B5

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superficial CO2 laser resurfacing (Experimental): The tested product and comparators are applied twice daily from Day2 to Day18 (except Sundays Day7 and Day14). Each subject receives a total of 30 applications of each tested product.
  Interventions: Other: superficial CO2 laser resurfacing
- Laser untreated side (Active Comparator): The tested product and comparators are applied twice daily from Day2 to Day18 (except Sundays Day7 and Day14). Each subject receives a total of 30 applications of each tested product.
  Interventions: Other: Laser untreated side

INTERVENTIONS:
Other: superficial CO2 laser resurfacing — Application of the tested product and comparators on the laser treated side of the back
  Arms: superficial CO2 laser resurfacing
Other: Laser untreated side — Application of the tested product and comparators on the laser untreated (control) side of the back
  Arms: Laser untreated side

SUMMARY:
This monocentric, double-blinded, randomized with intra-individual comparisons study is an interventional cosmetic study.

The objective is to evaluate the effectiveness of a new formulation on the re-epithelialization kinetic after superficial CO2 laser dermabrasion in comparison to an untreated area.

DETAILED DESCRIPTION:
This clinical trial is conducted in accordance with the protocol, the Helsinki declaration (1964) and subsequent amendments, and the International Council on Harmonisation (ICH) Good Clinical Practice (GCP), and in compliance with applicable regulatory requirements.

Statistical method: analysis will be performed using R software version 4.0.2. or higher. All statistical tests will be two-sided and at the 5% level of significance. Normality tests will be at the 1% level of significance (Shapiro-Wilk). All efficacy evaluation will be done on the Per Protocol Set.

The categorical variables are summarized by frequency and percentage for each response category (N, %). The continuous variables are summarized using means, medians, minimum, maximum, and standard deviations for the data collected at each visit.

Sample size determination: A number of 22 subjects would allow to detect a significant difference of at least of 2 days for complete re-epithelialization score between the treated and untreated areas with a power of 91% at a risk alpha of 0.05 and assuming a common standard deviation of ±2.7 days. Twenty-five (25) subjects will be included in the study to take into account possible dropouts.

ELIGIBILITY:
Inclusion Criteria:

* phototype II and III on the Fitzpatrick scale
* subjects with normal clinical examination and medical history compatible with the study

Exclusion Criteria:

* subject with underlying pathology that may interfere with the interpretation of the study results (dermatological history of psoriasis, eczema, urticaria... or suspicion/history of allergies to cosmetics), skin abnormality (scars, excessive hair growth, tattoos...) in the test areas (back, midline), systemic pathology
* subject with excessive exposure to natural (sun) or artificial (tanning salon) ultraviolet light (UV) 4 weeks prior to the initial visit or who anticipates such exposure during the study
* subject who has taken systemic treatment for more than 5 days in the month prior to inclusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
wound healing assessment by the Investigator (number of days for complete re-epithelialization) | from baseline to Day19
  assessment on a 6-point scale: 0 (No healing); 1 (Weak healing: <25% of the lesion area); 2 (Partial healing: between 25 and 50% of the lesion area); 3 (Significant healing: between 50 and 75% of the lesion area); 4 (Almost complete healing: >75% of the lesion area); 5 (Complete healing).

SECONDARY OUTCOMES:
wound healing assessment by the Investigator (number of days for 25%, 50% and 75% re-epithelialization) | from baseline to Day19
  assessment on a 6-point scale: 0 (No healing); 1 (Weak healing: <25% of the lesion area); 2 (Partial healing: between 25 and 50% of the lesion area); 3 (Significant healing: between 50 and 75% of the lesion area); 4 (Almost complete healing: >75% of the lesion area); 5 (Complete healing).

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Queille-Roussel, Principal Investigator — Centre de Pharmacologie Clinique Applique a la Dermatologie
Locations (1):
- CPCAD, Nice, France